CLINICAL TRIAL: NCT06648369
Title: Maximal Medical Treatment of Intracerebral Haemorrhage Pilot Trial - MAX-ICH Pilot Trial
Acronym: MAX-ICH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MAX-ICH pilot trial
Record Dates: First submitted 2024-08-20; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Intra Cerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Single-center, randomized-controlled (2:1), two-arm parallel group, open treatment, blinded endpoint clinical trial (PROBE)
Who Masked: Outcomes Assessor
Masking Description: Blinded Endpoint Assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (usual care) (Other): Control group is treated according to local standard of care
  Interventions: Other: Standard of care
- Experimental arm (MAX-ICH care bundle) (Experimental): Experimental group is treated according MAX-ICH care bundle
  Interventions: Other: MAX-ICH care bundle

INTERVENTIONS:
Other: MAX-ICH care bundle — The MAX-ICH care bundle is a comprehensive treatment approach for intracerebral hemorrhage (ICH). Patients receive 72 hours of care in a high-dependency unit like an ICU or hyperacute stroke unit. Intensive blood pressure control is used if systolic blood pressure exceeds 140mmHg, with rapid reduction to below 140mmHg within 60 minutes, and maintenance at or above 110mmHg for at least 75% of the time, with variability kept under 20%. The protocol includes rapid reversal of anticoagulation within 60 minutes, administration of tranexamic acid (1g bolus within 60 minutes, followed by 1g over 8 hours), and neurosurgical evaluation within 60 minutes. Additionally, family counseling is provided to avoid Do-Not-Resuscitate orders during the first 72 hours.
  Arms: Experimental arm (MAX-ICH care bundle)
Other: Standard of care — The control group will be treated according to the hospital's standard protocol for patients with spontaneous intracerebral hemorrhage, based on the guidelines of the European Stroke Organisation (ESO). The ESO develops evidence-based recommendations for the optimal care of stroke patients. The recommended immediate measures include: immediate stabilization and assessment, blood pressure control and reduction, brain imaging, surgical intervention for large hemorrhages, coagulation control, and monitoring of intracranial pressure. The specific application of these measures varies depending on the hospital and the treating physicians.
  Arms: Control arm (usual care)

SUMMARY:
The MAX-ICH pilot trial is a phase-II study aimed at assessing the feasibility and safety of a comprehensive care bundle for patients with intracerebral hemorrhage (ICH). This "maximal medical treatment" approach combines advanced interventions like intensive blood pressure control, rapid anticoagulation reversal, and tranexamic acid administration to potentially improve outcomes. The primary objective is to evaluate recruitment feasibility over 12 months, while secondary objectives include protocol adherence, safety monitoring, and the exploration of clinical outcomes. The study focuses on the critical first 72 hours of care to determine if this approach can be effectively implemented in clinical practice.

DETAILED DESCRIPTION:
The MAX-ICH pilot trial is a monocentric, phase-II study designed to evaluate the feasibility and safety of a "maximal medical treatment" care bundle for patients suffering from intracerebral hemorrhage (ICH). ICH is a condition with a notably high rate of mortality and morbidity, and this trial aims to improve outcomes for these patients by utilizing a comprehensive approach to their treatment. Previous clinical trials concentrated on single interventions, such as blood pressure control and the administration of tranexamic acid (TXA) therapy. While these interventions did not achieve their primary efficacy outcomes, they did demonstrate beneficial effects on secondary measures like reducing hematoma expansion and early mortality. The current study builds on this prior research by integrating advanced interventions into a unified and comprehensive care bundle, termed MAX-ICH, with the goal of potentially enhancing patient outcomes.

The primary objective of the trial is to demonstrate the feasibility of recruiting patients within a 12-month period. In addition to this, secondary objectives include assessing the technical feasibility of protocol adherence, targeting a compliance rate of at least 70%. The study will also monitor safety by tracking major adverse cardiovascular events (MACE) and explore a range of clinical outcomes, treatment metrics, and differences between the experimental group receiving the MAX-ICH care bundle and those receiving standard care.

The MAX-ICH care bundle consists of several key components designed to deliver intensive and timely care. Patients will receive 72 hours of treatment in a high-dependency unit, ensuring continuous monitoring and rapid responses to any changes in their condition. Intensive blood pressure control will be implemented through intra-arterial monitoring to maintain stability. If a patient is on anticoagulant therapy, the care bundle mandates rapid reversal of anticoagulation within 60 minutes of presentation. Similarly, tranexamic acid will be administered within 60 minutes, helping to mitigate further hemorrhage. Neurosurgical evaluation will also be conducted within 60 minutes to determine if surgical intervention is warranted. Additionally, counseling will be provided to avoid placing Do-Not-Resuscitate (DNR) orders during the critical first 72 hours, allowing time for the intensive interventions to take effect.

Ultimately, this study aims to determine whether the MAX-ICH care bundle can be feasibly implemented in clinical practice and whether its structured, intensive approach within the first 72 hours of care can lead to improved outcomes for patients with ICH.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic imaging proven diagnosis of non-traumatic ICH
* Vascular imaging (MR-/CT-angiogram or DSA) on admission to rule out high suspicion of macrovascular bleeding source
* Enrolment no later than 6 hours of symptom onset
* Age >18 years, no upper age limit
* Informed consent as documented by signature or fulfilling the criteria for emergency consent/ deferral consent

Exclusion Criteria:

* Palliative care/comfort therapy decision in the emergency department
* ICH due to trauma (major head trauma <24 hours of symptom onset causing loss of consciousness and thought to be sufficient to have caused the intracerebral bleeding)
* High suspicion of ICH due to arteriovenous malformation (AVM), aneurysm or sinus-venous-thrombosis confirmed by neuroimaging, brain tumor, vasculitis, RCVS/PRES or system disease (liver disease, inherit coagulopathy)
* Severe ICH (haematoma volume >60ml or GCS <8)
* Haematoma evacuation or decompressive craniectomy within 72 hours planned or highly likely (isolated EVD is not an exclusion criterion)
* Severe pre-morbid disability [modified Rankin scale (mRS) is ≥4]
* Contraindication against the use of tranexamic acid
* Active participation in another drug or devices trial concurrently
* Female patient that are either pregnant or breastfeeding
* Contraindications against Clevidipine (allergy to soja, lipid metabolism defect or known severe aortic stenosis)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 12 months
  Recruitment rate at 12 months

SECONDARY OUTCOMES:
Technical feasibility | 12 months
  ≥70% compliance with MAX-ICH care bundle at 72 hours (experimental group only). Full compliance is defined as all 6 criteria of the MAX-ICH care bundle (for details see study intervention) are fulfilled. After the 12 months recruitment period the percentage of patients for which full compliance at 72h afer randomization to the care bundle group was achieved will be determined.
Major Adverse Cardiovascular Events | 30 days
  MACE within the first 30 days (i.e. Death, acute coronary syndrome (ACS) or myocardial infarction (MI), deep vein thrombosis (DVT), Pulmonary embolism (PE), VTE (combined DVT/PE), Ischaemic stroke)
Radiological outcomes | 24 hours
  Haematoma expansion at 24 hours
Radiological outcomes | 72 hours
  Presence and number of new lesions on DWI at 72 hours
Radiological outcomes | 72 hours
  Absolute and relative PHE volume on FLAIR at 72 hours
Clinical outcomes | 24 hours
  Mortality at 24 hours
Clinical Outcome | 24 hours
  Early functional outcome (Modified Rankin Scale (mRS 0-6, no symptoms - death)) at 24 hours
Clinical Outcome | 24 hours
  Early functional outcome (National Institutes of Health Stroke Scale (NIHSS 0-42, no symptoms - severe stroke)) at 24 hours
Clinical outcomes | 72 hours
  Mortality at 72 hours
Clinical Outcome | 72 hours
  Functional outcome (Modified Rankin Scale (mRS 0-6, no symptoms - death)) at 72 hours
Clinical Outcome | 72 hours
  Functional outcome National Institutes of Health Stroke Scale (NIHSS 0-42, no symptoms - severe stroke)) at 72 hours
Clinical outcomes | 3 months
  Mortality at 3 months
Clinical Outcome | 3 months
  Functional outcome (Modified Rankin Scale (mRS 0-6, no symptoms - death)) at 3 months
Clinical outcomes | 6 months
  Mortality at 6 months
Clinical Outcome | 6 months
  Functional outcome (Modified Rankin Scale (mRS 0-6, no symptoms - death)) at 6 months
Quality of blood pressure control | 60 min
  Rapidity (<60minutes from randomization to reach target blood pressure level)
Quality of blood pressure control | 72 hours
  Sustainability (≥70% of time within target blood pressure level during treatment)
Quality of blood pressure control | 72 hours
  Variability (<20% variability of blood pressure level during treatment)
Quality of blood pressure control | 72 hours
  Hypotensive episodes (time below lower threshold)
Between group differences | 72 hours
  Treatment delivery (% of patients receiving treatment)
Between group differences | 72 hours
  Metrics (time to treatment, time to target)

CONTACTS AND LOCATIONS:
Overall Officials: David J Seiffge, Prof. Dr. med., Principal Investigator — Department for Neurology, Inselspital, University Hospital Bern
Locations (1):
- Inselspital, University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Not shared